CLINICAL TRIAL: NCT01446432
Title: A Prospective Study to Validate Two New Patient Reported Outcome Measures for Dupuytren's Disease in Patients Treated With XIAFLEX
Brief Title: Validation of Two New Questionnaires for Dupuytren's Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Robert Hotchkiss (Other)
Collaborators: Auxilium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Robert Hotchkiss, MD, Hospital for Special Surgery, New York
Organization: Hospital for Special Surgery, New York (Other)
Other Study IDs: 11011
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Dupuytren's Disease
Keywords: Dupuytren's Contracture
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A study to validate two newly developed questionnaires for Dupuytren's Disease. The objective is to develop a patient specific outcomes tool for Dupuytren's Disease. While there are standard and validated questionnaire instruments used to measure health related quality of life and function, they do not address patient specific issues. The investigators will also pilot a treatment/disease specific satisfaction questionnaire for Xiaflex use for Dupuytren's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of Dupuytren's Disease in at least one finger
* Patients will be 35 years of age or older
* Patients will be able to read, speak, and understand English
* Patients will be able to provide voluntary written consent to participate

Exclusion Criteria:

* Female patients who are nursing or pregnant, or plan to become pregnant during the treatment phase.
* Patient has a chronic muscular, neurological or neuromuscular disorder that affects the hands.
* Patient has a known allergy to collagenase or any other excipient of XIAFLEX.
* Patient has received any collagenase treatments before the first dose of XIAFLEX.
* Any history of or current medical condition which in the investigator's opinion would make the subject unsuitable for enrollment in the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment with XIAFLEX for Dupuytren's Disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
QuickDASH (Disability of the Arm, Shoulder, and Hand) | 30 day follow up

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Hotchkiss, MD, Principal Investigator — Hosptial for Special Surgery
Locations (1):
- Hospital For Special Surgery, New York, New York, United States